CLINICAL TRIAL: NCT04271839
Title: Open Randomized Low Interventional Clinical Trial to Compare Efficiency in Control Symptoms Between Fluticasone Propionate/Formoterol K-haler (Medium Strength) vs High Strength ICS/LABA in the Treatment of Patients With Persistent Asthma
Brief Title: Efficiency Control of Fluticasone/Formoterol K-haler (Medium Strength) vs ICS/LABA (High Strength) in Asthma Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The trial has been terminated early due to the SARS-CoV-2 pandemic.
Sponsor: Mundipharma Pharmaceuticals S.L. (Industry)
Collaborators: Alpha Bioresearch S.L. (Other); Dynamic Solutions (Industry)
Responsible Party: Principal Investigator, Rubén Lesmes Escudero, Clinical Professor, Mundipharma Pharmaceuticals S.L.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EffICIENCY
Record Dates: First submitted 2020-02-11; First posted 2020-02-17 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-02

CONDITIONS: Persistent Asthma
MeSH Terms: interventions — Fluticasone; Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluticasone/formoterol k-haler (medium strength) (Experimental): In this arm, uncontrolled patients who arrive at the consultation with their fixed combination of ICs (Inhaled CorticosteroidS) / LABA (Long-Acting Beta2-Agonist) (medium strength) will change their treatment to Fluticasone / formoterol k-haler (medium strength)
  Interventions: Combination Product: fluticasone/formoterol k-haler (medium strength)
- Standard of Care (SoC) (Active Comparator): In this arm, uncontrolled patients arriving at the consultation with their fixed combination of ICs / LABA (medium strength) will change their treatment to the same fixed combination of ICs / LABA (high strength)
  Interventions: Combination Product: Standard of care (ICs/LABA high strength)

INTERVENTIONS:
Combination Product: fluticasone/formoterol k-haler (medium strength) — 2 inhalations every 12 hours
  Other Names: No other interventions
  Arms: Fluticasone/formoterol k-haler (medium strength)
Combination Product: Standard of care (ICs/LABA high strength) — Depend of the ICs/LABA combination
  Other Names: No other interventions
  Arms: Standard of Care (SoC)

SUMMARY:
Clinical trial to demonstrate whether, in patients with moderate asthma, to treat with IC / LABA a medium dose, but not controlled, to achieve a similar degree of control by making a progressive increase of that treatment (CI / LABA a high dose) versus switching to fluticasone / Formoterol K-Haler at medium dose, under conditions of usual clinical practice.

DETAILED DESCRIPTION:
Asthma is a common chronic respiratory disease that affects about 300 million people worldwide. Although knowledge about asthma and its treatment has improved over the past decade, morbidity and mortality remain considerable.

Inhaled therapy is the treatment of choice in persistent asthma. Lower doses of drug are used that maximize the therapeutic effect and minimize side effects.

Inhaled therapy is administered primarily through inhalers. The goal is to deliver the maximum amount of medication to your therapeutic target in the lungs → lung deposit Each inhaler offers a different lung deposit figure (data in ideal conditions). However, asthma control also depends on other factors (inhalation technique, adhesion, asthma severity, drug dose, etc.).

The K-haler® inhaler device has obtained a high lung deposit (≈45% of the emitted dose) and an easy-to-use device.

In general, the rest of the CI / LABA inhalers offer lower deposit figures. They are between ≈10-40% of the dose.

Taking into account all that has been said in the introduction section, it has been decided to design this low-intervention clinical trial, to verify whether, those technical benefits of K-haler®, control asthma in a similar way using lower doses of IC .

If these hypotheses were confirmed, it would allow for an effective therapeutic option in the control of asthma using a lower therapeutic dose, saving IC and a lower probability of producing side effects.

Demonstrate whether, in patients with moderate asthma, to treat with IC / LABA a medium dose, but not controlled, to achieve a similar degree of control by making a progressive increase of that treatment (CI / LABA a high dose) versus switching to fluticasone / Formoterol K-Haler at medium dose, under conditions of usual clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Age > or = 18 years.
2. Objective diagnosis of asthma (according to GEMA 4.4) (Guía Española de Manejo del Asma)
3. Patients in treatment with a stable average dose of IC in a fixed dose combination of IC / LABA *, without changes in the dose or in the inhaler, during the 3 months prior to inclusion, in accordance with its approved indication and Data sheet. * Except for K-Haler®
4. Patients who need, according to medical criteria, a dose increase of IC in the current fixed IC / LABA combination.
5. Inhalation technique: no critical errors with the current inhaler after training.
6. Patient with uncontrolled asthma with an ACQ> 0.75 points (partially controlled or poorly controlled asthma).
7. Informed consent in signed writing.

Exclusion Criteria:

1. Diagnosis of other respiratory pathology other than asthma (clinically relevant bronchiectasis, pulmonary fibrosis, COPD (Chronic Obstructive Pulmonary Disease) and others at the discretion of the investigator).
2. ≥1 severe exacerbation (require the use of systemic corticosteroids - oral, suspension or injection - or increasing the dose of maintenance therapy for at least 3 days, or hospitalization or emergency room visits due to asthma requiring the use of systemic corticosteroids) in the last month or ≥3 in the previous 12 months.
3. Pregnancy or probability of being pregnant during the study.
4. Patient who, at the discretion of the investigator, does not have the capacity to complete the questionnaires.
5. Patient under treatment with monoclonal antibodies during the study.
6. Patient in another clinical trial.
7. Patient who has received an experimental drug in the last 30 days (12 weeks if it is a systemic steroid).
8. Do not use a MART (MAintenance and Reliever Therapy) strategy within 3 months prior to inclusion or during the trial
9. Patient in IC / LABA treatment according to MART strategy (Maintenance and Rescue).
10. Any contraindication expressed in the CI / LABA data sheet used.
11. Patient with poor adherence (TAI-10 ≤ 45)
12. Patients using an inhalation chamber
13. Patients with an index of Packages / year> 10

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Control of asthma | 24 weeks
  The control of asthma in patients with persistent asthma will be measured by scoring the ACQ-7 questionnaire (Asthma Control Questionnaire): Well controlled: ≤ 0.75, Partially controlled: from 0.75 to 1.50, Poorly controlled:> 1.50

SECONDARY OUTCOMES:
Degree of asthma control according to GINA (Global Initiative for Asthma) questionnaire of four questions | 24 weeks
  Well Controlled (negative answer in the 4 questions), Partially controlled (affirmative answer in 1 or 2 of the answers), Uncontrolled (affirmative answer in 3 or 4 of the answers)
Success in asthma treatment | 24 weeks
  Defined as asthma patients who progress from poorly controlled asthma to partially or well controlled asthma, or from partially controlled asthma to controlled asthma, with no change in baseline asthma treatment after randomization
  Measured by scoring the ACQ-7 questionnaire: Well controlled: ≤ 0.75, Partially controlled: from 0.75 to 1.50, Poorly controlled:> 1.50
Adherence to treatment | 24 weeks
  Through TAI-12 questionnaire (Erratic Total Score 1-5 items, Deliberate Total Score 6-10 items, Unconscious Total Score 11-12 items) And through electronic prescription (if the amount of medication withdrawn in pharmacy matches that prescribed by the doctor)
Critical errors with the inhaler | 24 weeks
  Number of critical errors
Patient satisfaction with the inhaler | 24 weeks
  Through the FSI-10 (Feeling of Satisfaction with Inhaler) questionnaire (It consists of 10 questions, each with 5 response options on a 5-step Likert scale ("a lot", "a lot", "something", "little" and "very little") scored, respectively, from 5 to 1 (score total: 50). It evaluates the degree of patient satisfaction with the inhalation device and includes items related to comfort, difficulty, transportability and use.)
Quality of Life of the patient | 24 weeks
  Through Mini-AQLQ (Mini Asthma Quality of Life Questionnaire) questionnaire: This 15-item questionnaire is a short version of the complete 32-item questionnaire, but constitutes of the same 4 domains: symptoms, environment, emotions, activities, and covering a 2 week period. Scores range from 0-6 (lower is worse). The mini-AQLQ score is calculated as the average of domain items. The minimum clinically important difference is 0.5.
  This version has been developed to meet the needs of long-term monitoring, where efficiency may take precedent over precision of measurement
Severe asthmatic exacerbations | 24 weeks
  Number severe asthmatic exacerbations (require the use of systemic corticosteroids - oral, suspension or injection - or the increase in the dose of maintenance therapy for at least 3 days, or hospitalization or visits to the emergency room due to asthma that requires the use of systemic corticosteroids)
Forced Expiratory Volume at first second (FEV1) | 24 weeks
  Using the FEV1 score of the patient's spirometry
Forced Vital Capacity (FVC) | 24 weeks
  Using the FVC score of the patient's spirometry
FEV1 / FVC ratio | 24 weeks
  Using the FEV1 and FVC score of the patient's spirometry
Safety of the drug in investigation. | 24 weeks
  Type and incidence of adverse reactions

CONTACTS AND LOCATIONS:
Overall Officials: José Luis Velasco Garrido, MD, Study Director — Hospital Virgen de la Victoria; Javier Domínguez Ortega, MD, Study Director — Hospital La Paz; Patricia García Sidro, MD, Principal Investigator — Hospital La plana; Ernesto Enrique Miranda, MD, Principal Investigator — Hospital General de Castellón; Ana Gómez-Bastero Fernández, MD, Principal Investigator — Hospital Universitario Virgen Macarena; Alicia Padilla Galo, MD, Principal Investigator — Hospital Costa del Sol; Fernando Florido López, MD, Principal Investigator — Hospital San Cecilio; Joaquín Quiralte Enriquez, MD, Principal Investigator — Hospital Virgen del Rocío; Antolín López Viña, MD, Principal Investigator — Hospital Puerta de Hierro; Carlos Almonacid Sánchez, MD, Principal Investigator — Hospital Universitario Ramon y Cajal; María del Mar Gandolfo Cano, MD, Principal Investigator — Hospital de Fuenlabrada; Paula López González, MD, Principal Investigator — Hospital Infanta Leonor; Blanca Requejo Mañana, MD, Principal Investigator — Hospital Central de Asturias; Ana Pando Sandoval, MD, Principal Investigator — Hospital Central de Asturias; Carlos Martínez Rivera, MD, Principal Investigator — Germans Trias i Pujol Hospital; Xavier Muñoz Gall, MD, Principal Investigator — Hospital Vall d'Hebrón; Gaspar Dalmau Duch, MD, Principal Investigator — Hospital Joan XXIII; Luis Alejandro Pérez de Llano, MD, Principal Investigator — Hospital Lucus Augusti; Abel Pallarés Sanmartín, MD, Principal Investigator — Complejo Hospitalario Universitario de Vigo; Vanesa García Paz, MD, Principal Investigator — Complejo Hospitalario Universitario de Santiago de Compostela; Francisco Javier Callejas González, MD, Principal Investigator — Hospital del Perpetuo Socorro de Albacete; Patricia Prieto Montaño, MD, Principal Investigator — Hospital del Perpetuo Socorro de Albacete; Ana Tabar Purroy, MD, Principal Investigator — Complejo Hospitalario de Navarra